CLINICAL TRIAL: NCT04609852
Title: A Randomized, Single-Blind, Placebo-Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of E8001 in Healthy Male Subjects
Brief Title: A Study to Assess the Safety and Tolerability of E8001 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: E8001-J081-001
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-03

CONDITIONS: Healthy Volunteers
Keywords: Healthy Participants; E8001

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1: E8001 or Placebo (Experimental): Participants will receive specified dose of E8001 or placebo (isotonic sodium chloride solution), infusion, intravenously, once on Day 1.
  Interventions: Drug: E8001; Drug: Placebo
- Cohort 2: E8001 or Placebo (Experimental): Participants will receive specified dose of E8001 or placebo (isotonic sodium chloride solution), infusion, intravenously, once on Day 1.
  Interventions: Drug: E8001; Drug: Placebo
- Cohort 3: E8001 or Placebo (Experimental): Participants will receive specified dose of E8001 or placebo (isotonic sodium chloride solution), infusion, intravenously, once on Day 1.
  Interventions: Drug: E8001; Drug: Placebo
- Cohort 4: E8001 or Placebo (Experimental): Participants will receive specified dose of E8001 or placebo (isotonic sodium chloride solution), infusion, intravenously, once on Day 1.
  Interventions: Drug: E8001; Drug: Placebo

INTERVENTIONS:
Drug: E8001 — Intravenous infusion.
Drug: Placebo — Intravenous infusion.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (PK) of E8001 of single ascending dose intravenous infusions in healthy male participants.

ELIGIBILITY:
Inclusion Criteria

1. Non-smoking, age greater than or equal to (>=) 20 years and less than or equal to (<=) 55 years old adult male at the time of informed consent. To be considered non-smokers, participants must have discontinued smoking for at least 4 weeks before dosing
2. Body mass index (BMI) >=18.5 and less than (<) 25.0 kilogram per square meter (kg/m˄2) at Screening

Exclusion Criteria:

1. Males who have not had a successful vasectomy (confirmed azoospermia) or they and their female partners do not meet the criteria (that is, not of childbearing potential or practicing highly effective contraception throughout the study period or for 5 times the half-life of the study drug plus 90 days after study drug discontinuation). No sperm donation is allowed during the study period and for 5 times the half-life of the study drug plus 90 days after study drug discontinuation
2. Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks of dosing
3. History of meningococcal infection or pneumococcal infection
4. Evidence of disease that may influence the outcome of the study within 4 weeks before dosing; example- psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or participants who have a congenital abnormality in metabolism
5. Any history of gastrointestinal surgery that may affect PK profiles of E8001, example- hepatectomy, nephrectomy, and digestive organ resection at Screening
6. Any clinically abnormal symptom or organ impairment found by medical history at Screening, and physical examinations, vital signs, ECG finding, or laboratory test results that require medical treatment at Screening or Baseline
7. History of prolonged QT/QTc interval
8. History of left bundle branch block (LBBB)
9. History of myocardial infarction (MI) or active ischemic heart disease (IHD)
10. History of clinically significant arrhythmia or uncontrolled arrhythmia
11. Active viral hepatitis (A, B or C) and syphilis as demonstrated by positive serology at Screening
12. History of drug or alcohol dependency or abuse, or those who have a positive drug test at Screening or Baseline
13. Liver function test with following values at Screening or Baseline:

    1. aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), or gamma glutamyl transpeptidase (GGT): greater than (>) upper limit of normal (ULN)
    2. direct bilirubin or total bilirubin: >1.5*ULN

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Screening up to Day 180 (approximately 292 days)
  Safety assessments will consist of monitoring and recording all adverse events (AEs) and SAEs; regular monitoring of clinical laboratory parameters; and periodic measurement of vital signs and 12-lead electrocardiogram (ECG), body weight and physical examinations.
Cmax: Maximum Observed Plasma Concentration for E8001 | Day 1: 0-168 hours
Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for E8001 | Day 1: 0-168 hours
AUC(0-t): Area Under the Concentration-time Curve From Zero (Pre-dose) to Time of Last Quantifiable Concentration for E8001 | Day 1: 0-168 hours
T1/2: Terminal Elimination Phase Half-life for E8001 | Day 1: 0-168 hours
CL: Total Clearance for E8001 | Day 1: 0-168 hours
Vss: Volume of Distribution at Steady State for E8001 | Day 1: 0-168 hours

SECONDARY OUTCOMES:
Change From Baseline in Corrected QT (QTc) Interval | Day 1: 0-24 hours
  To assess the effect of E8001 on ventricular repolarization by assessing the QTc interval corrected by the Fridericia formula (QTcF).

CONTACTS AND LOCATIONS:
Locations (1):
- Eisai Trial Site #1, Minatoku, Japan

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

REFERENCES:
- [Derived] Ishigooka H, Katsumata H, Saiga K, Tokita D, Motoi S, Matsui C, Suzuki Y, Tomimatsu A, Nakatani T, Kuboi Y, Yamakawa T, Ikeda T, Ishii R, Imai T, Takagi T, Tanabe K. Novel Complement C5 Small-interfering RNA Lipid Nanoparticle Prolongs Graft Survival in a Hypersensitized Rat Kidney Transplant Model. Transplantation. 2022 Dec 1;106(12):2338-2347. doi: 10.1097/TP.0000000000004207. Epub 2022 Nov 22. PMID 35749284